CLINICAL TRIAL: NCT06544213
Title: A Randomized Controlled Study on 24 Healthy Male Volunteers Evaluating the Effects of Centrifugation and Exercise to Prevent the Deconditioning Induced by 60 Days of Head-down Bedrest Used as a Ground-based Model to Mimic Weightlessness.
Brief Title: A 60 Days Head Down Tilt Bedrest With Artificial Gravity and Cycling Exercise on 24 Healthy Male (BRACE)
Acronym: BRACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National d'Etudes Spatiales (Other Government)
Collaborators: European Space Agency (Other); MEDES - IMPS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-242; 2022-A02074-39 (Other: IDRCB)
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Simulated Microgravity by Head Down Tilt Bedrest; Weightlessness
Keywords: Simulation of microgravity; Weightlessness; Artificial Gravity; Bedrest; Countermeasure
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Volunteers are divided in three groups (8 volunteers each), one control group, one group with supine bike as countermeasure, one group with artificial gravity and supine bike as countermeasure
Masking Description: Participants and investigators are aware of the groups distribution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): Control group does not receive any countermeasure program during the head down tilt phase.
  Interventions: Behavioral: Control Group
- Artificial Gravity and Supine Bike (Experimental): The volunteers in this group receive countermeasure exercises during the head down tilt phase.
  6 days over 7, they will perform a 30 minutes exercises on a supine bike (incremental steps) combined with artificial gravity generated with a short arm centrifuge.
  Interventions: Behavioral: Countermeasure AG-Bike
- Supine Bike (Experimental): The volunteers in this group receive countermeasure exercises during the head down tilt phase.
  6 days over 7, they will perform a 30 minutes exercises on a supine bike (incremental steps).
  Interventions: Behavioral: Countermeasure Supine Bike

INTERVENTIONS:
Behavioral: Control Group — 60 days of strict head down tilt bed rest at all time. No countermeasure program is performed.
  Arms: Control Group
Behavioral: Countermeasure Supine Bike — 60 days of strict head down tilt bed rest at all time. The exercise starts at 40% of VO2max for 5 minutes, followed by a series of 2-minute high- and low-intensity intervals for 20 minutes. 2-minute high-intensity intervals are at 65% VO2max, 70% VO2max, 80% VO2max, 80% VO2max, 70% VO2max and 65% VO2max. 2-minute low-intensity intervals are at 40% VO2max. 3 minutes at 40% of VO2max will end the exercise.
  VO2max is measured for each volunteer in supine position.
  Arms: Supine Bike
Behavioral: Countermeasure AG-Bike — 60 days of strict head down tilt bed rest at all time. The exercise starts at 40% of VO2max for 5 minutes, followed by a series of 2-minute high- and low-intensity intervals for 20 minutes. 2-minute high-intensity intervals are at 65% VO2max, 70% VO2max, 80% VO2max, 80% VO2max, 70% VO2max and 65% VO2max. 2-minute low-intensity intervals are at 40% VO2max. 3 minutes at 40% of VO2max will end the exercise.
  VO2max is measured for each volunteer in supine position.
  The supine bike exercise is performed in a short arm centrifuge in rotation. Volunteers will start pedalling and the centrifuge will start at 0.15 Gz less than individual's threshold.
  Every 4 minutes thereafter, the AG will be increased by 0.15 Gz, synchronized with the ramping up of cycle ergometer interval intensity. The AG will increase only up to 70 % of their tolerance level,.
  It will then decrease by 0.15 Gz every 4 minutes, and until the 30-minute exercise is completed.
  Arms: Artificial Gravity and Supine Bike

SUMMARY:
The objective of this study is to investigate whether a cycling exercise coupled with artificial gravity via a short-arm human centrifuge helps to prevent and / or reduce the deleterious effects induced by 60 days of anti-orthostatic bedrest.

The secondary objective is to investigate whether the combination of a supine cycling exercise with artificial gravity is more effective than the same supine cycling exercise alone in preventing or reducing the effects of head-down bedrest.

During a randomized, 60 day bed rest study, in 24 healthy male adults, the two following aims will be undertaken:

* Fourteen scientific protocols will assess the changes in the cardiovascular, metabolic, musculoskeletal, neuro-sensorial, haematological, and immunological systems.
* In the above-mentioned systems, the comparative potential beneficial effects of the two countermeasure protocols will also be investigated by the scientific protocols and bedrest standard measurements (BSM).

DETAILED DESCRIPTION:
Space flights have shown the possibilities and limitations of human adaptation to space. For the last 60 years, results have shown that the space environment and microgravity in particular, cause changes that may affect the performance of astronauts. These physiological changes are now better known: prolonged exposure to weightlessness can lead to significant loss of bone and muscle mass, strength, cardiovascular and sensory-motor deconditioning, immune, hormonal and metabolic changes .

Moreover, recently a new suite of physiological adaptations and consequences of space flight has been acknowledged. Indeed, after long flights, some astronauts present persistent ophthalmologic changes, mostly a hyperopic shift, an increase in optic nerve sheath diameter and occasionally a papillary oedema now defined by National Aeronautics and Space Administration (NASA) as Spaceflight-Associated Neuro-ocular Syndrome (SANS). Some of these vision changes remain unresolved for years post-flight. This phenomenon has most likely existed since the beginning of human space flight but is just recently being recognized as a major consequence of adaptation to microgravity.

Overall, spaceflight induces physiological multi-system deconditioning which may impact astronauts' efficiency and create difficulties upon their return to normal gravity. Understanding the underlying mechanisms of these processes and developing efficient countermeasures to prevent, limit or reverse this deconditioning remain important challenges and major priorities for manned space programs.

The space agencies are actively engaged in studying the physiological adaptation to space environment through studies on board the International Space Station (ISS) but also on the ground. Indeed, considering the limited number of flight opportunities, the difficulties related to the performance of in-flight experiments (operational constraints for astronauts, limited capabilities of in-flight biomedical devices), ground-based experiments simulating the effects of weightlessness are used to better understand the mechanisms of physiological adaptation, design and validate the countermeasures.

Different methods are used to simulate microgravity on Earth. However, two approaches, -6° head-down bed rest (HDBR) and dry immersion (DI) have provided possibilities for long-term exposures with findings closest to those seen with a weightless state. They produce changes in body composition (including body fluid redistribution), cardiovascular and skeletal muscle characteristics that resemble the effects of microgravity. One of the advantages of the HDBR model is that it has now been used in a great number of studies internationally, and its effects have long been described and compared with those of microgravity and spaceflight. Long-term bedrest is the gold-standard method for studying the effects of weightlessness and to test countermeasures.

The HDBR, as the name implies, implicates a long (from several weeks to a year) stay in the supine position, the head tilted down by -6° from the horizontal plane. HDBR is the most frequently used ground-based simulation for gravitational unloading of the human body in western countries.

During human space missions, the current most effective countermeasure is physical exercise. However, it is both time-consuming and not completely satisfactory. One of the solutions for this is to combine physical exercise with artificial gravity, with the use of a short-arm human centrifuge (SAHC). This study proposes to test the effectiveness of a countermeasure protocol combining Artificial Gravity (AG) with a cycling exercise, and to compare it with only a cycling exercise, and with a complete lack of physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer (see below the description of medical tests and laboratory analysis performed at the selection visit)
* Aged 20 to 45 years
* No overweight nor excessive thinness with BMI (weight kg/ height m2) between 20 and 27 kg/m2
* Height between 158 and 190 cm
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination): in particular, free from any chronic disease or any acute infectious disease or cardiovascular, neurological, of the ear, nose, throat (especially orthostatic hypotension and vestibular disorders), orthopaedic or musculoskeletal disorders
* Good mental health: tests and psychological interview will be held by a specialist in extreme environment
* Fitness level assessment: 35 mL/min/kg < VO2max < 55 mL/min/kg
* Non active smokers
* No alcohol or drug dependence, and no medical treatment
* Covered by a Health Insurance System
* Having signed the information consent
* Free of any engagement during the study

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, neurological or ear, nose, throat disease, any chronic disease; any acute infectious disease. Particularly:
* Symptomatic orthostatic hypotension whatever the decrease in blood pressure, or asymptomatic postural hypotension defined by a decrease in systolic blood pressure equal to or greater than 20 mmHg within 3 minutes when changing from the supine to the standing position,
* Cardiac rhythm disorders,
* Hypertension,
* Chronic back pains,
* Vertebral fracture, scoliosis, or herniated disc,
* Glaucoma,
* Self-reported hearing problems,
* Vestibular disorders
* History of migraines,
* History of hiatus hernia or gastro-esophageal reflux,
* History of thyroid dysfunction, renal stones, diabetes,
* History of head trauma,
* Abnormal result for lower limbs echo-doppler,
* History of genetic muscle and bone diseases of any kind,
* Past records of thrombophlebitis, family history of thrombosis or positive response in thrombosis screening procedure (anti thrombin III, S-protein, C-protein, factor V Leiden mutation and the mutation 20210 of the prothrombin gene),
* Bone mineral density: T-score ≤ -1.5,
* Poor tolerance to blood sampling,
* Having given whole blood (more than 7 mL/kg) in a period of 8 weeks or less before the start of the experiment, or having given whole blood more than 2 times in the past year,
* Significant history of allergy, especially no dermatological or food allergy,
* Significant anomaly detected in the biological analysis,
* Positive reaction to any of the following tests: hepatitis A immunoglobulin, hepatitis B antigen, anti hepatitis C antibodies, anti Human Immunodeficiency Virus 1+2 antibodies,
* Vegetarian or vegan,
* Refusal to give permission to contact his general practitioner,
* Subject who, in the judgment of the investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development,
* Subject already participating or in the exclusion period of a clinical research,
* Subject who has received more than 4500 Euros within 12 months for being a research subject,
* Subject who cannot be contacted in case of emergency,
* Subject who had the two knees injured
* MRI contraindications
* History or active claustrophobia
* Osteosynthesis material, presence of metallic implants or any other contra-indication for MRI
* Vulnerable persons according to French law (L1121-5 to L1121-8) :
* Persons deprived of their liberty by an administrative or judicial decision
* Persons under involuntary psychiatric care
* Persons admitted in a health or social establishment for purposes other than research
* Minors
* Adults subject to legal protection (subject under guardianship or trusteeship) or unable to express their consent

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in orthostatic tolerance | At baseline and first day of recovery
  Orthostatic tolerance will be assessed during a tilt test combined with Lower Body Negative Pressure test (LBNP test)
Changes in peak aerobic power (VO2max test) | At baseline and end of head down tilt phase at week 10
  Exercise capacity wil be assessed by graded cycling on sitting ergometer until exhaustion
Changes in plasma volume | At baseline and end of head down tilt phase at week 10
  Plasma volume (L) will be assessed by the carbon monoxide-rebreathing method
Changes in serum bone formation markers | From baseline until the end of the volunteers' participation in the study at year 2
  Change in bone-specific Alkaline Phosphatase (bAP, µg/L) and procollagen type I N-terminal propeptide (P1NP, µg/L) will be assessed by chemiluminescence immunoassay
Change in serum bone resorption markers | From baseline until the end of the volunteers' participation in the study at year 2
  Change in C-terminal cross-linked telopeptide of type I collagen (CTx, pmol/L) and N-terminal cross-linked telopeptide of type I collagen (NTX, pmol/L) will be assessed by chemiluminescence immunoassay.
Changes in Resting Metabolic Rate (RMR) | At baseline and at recovery at week 12
  RMR will be measured by indirect calorimetry technique
Change in nitrogen balance | At baseline and at recovery at week 12
  Nitrogen balance is a measure of nitrogen input minus nitrogen output. Nitrogen intake is calculated with a nutrition software. Protein oxidation measured in the 24-Hour urine collection estimates nitrogen output.
Change in muscle strength | At baseline and at recovery at week 10
  Muscle strength will be assessed from single leg isometric maximal voluntary contraction on the knee extensors & flexors, the plantarflexors and dorsiflexors. The Isometric Torque will be measured in Nm. The peak of the three maximal attempts will be recorded for strength measures
Change in fat and lean body mass measured by dual energy x-ray absorptiometry (DEXA) | From baseline until the end of the volunteers' participation in the study at year 2
  Dual energy x-ray absorptiometry is a standard clinical technique to assess fat (g) and lean (g) body mass.
Change in walking balance | At baseline and at recovery at week 10
  Functional mobility test (such as sit and walk, heel to toe steps with eyes closed and open) will assess walking balance
Changes in jump performance | At baseline and at recovery at week 12
  Jump performance will be assessed on a platform and height of the jump will be evaluated
Change in standing balance | At baseline and at recovery at week 10
  Standing balance will be assessed by posturography eyes open and eyes closed on a platform covered with 12-cm thick medium density foam
Changes in leg muscle volume and fat | At baseline and at recovery at week 10
  MRI of the lower extremity will assess the degree of atrophy and changes in fat content in the musculature
Changes in bone density (by DEXA and High Resolution Peripheral Computed Tomography (HR-pQCT)) | From baseline until the end of the volunteers' participation in the study at year 2
  Bone density is measured at lumbar and hip level with DEXA and at tibia and radius level with HR-pQCT
Change in the optic nerve fibers thickness | At baseline and at recovery at week 12
  Thickness of the optic nerve fibers will be measured by Optical Coherence Tomography (OCT)
Change in intraocular pressure (IOP) | At baseline and at recovery at week 12
  IOP is measured with air tonometry
Change in visual acuity | At baseline and at recovery at week 12
  Far and near visual acuity are tested uncorrected, or if applicable with own correction with digital acuity system
Change in visual field | At baseline and at recovery at week 12
  Visual field measured by standard automated perimetry
Change in the anatomical characteristics of the eye (optical biometry) | At baseline and at recovery at week 12
  Optical biometry measured by partial coherence interferometry
Change in the central corneal thickness | At baseline and at recovery at week 12
  Central corneal thickness on a single point on the cornea measured by Ultrasonic pachymetry
Change in the retina by non-mydriatic fundus retinography | At baseline and at recovery at week 12
  Non-mydriatic fundus retinography allows a fundus photography to be taken and thus a color image of the papilla, retinal vessels and macula
Change in the cornea topography | At baseline and at recovery at week 12
  Cornea topography measured by corneal topography equipment (like Pentacam). The elevation topography allows the mapping of the anterior and posterior surface of the cornea.
Change in motion sickness susceptibility | At baseline and at recovery at week 12
  Assessed by the Motion Sickness Susceptibility Questionnaire Short form (MSSQ-Short). MSSQ-Short scores possible range from minimum 0 to maximum 54, the maximum being unlikely. Higher scores means a higher motion sickness susceptibility
Change in fluid shift distribution towards the cardiac and cephalic region | At baseline and until year 1
  The consequences of the fluid shift on the cardiac and cephalic area will be assessed by quantifying the right and left Jugular veins volumes (mL), as well as the left ventricle diastolic/systolic volumes (mL) by ultrasound.
Change in mood | At baseline and until week 12
  Change in mood is assessed using the Profile of Mood States (POMS) questionnaire. POMS questionnaire gives 6 measures of mood:
  Tension/anxiety, Depression, Anger/hostility Dynamism, Fatigue, Confusion A Total Mood Disturbance (TMD) score is calculated by summing the totals for the negative subscales (tension, depression, fatigue, confusion, anger) and then subtracting the totals for the positive subscale (vigor /esteem-related affect).
Change in affective states | At baseline and until week 12
  Positive and Negative Schedule (PANAS) questionnaire will be used to assess the intensity of positive and negative affective states. PANAS self-report questionnaire consists of two 10-item scales to measure both positive and negative affects
  Each item is rated on a five-point Likert Scale, ranging from 1 = Not at all to 5 = Extremely, to measure the extent to which the affect has been experienced in a specified time frame.
  Positive affects: scores can range from 10 - 50 with higher scores representing higher levels of positive affect.
  Negative affects: scores can range from 10 - 50 with higher scores representing higher levels of negative affect.
Change in sleep quality | At baseline and until week 12
  Pittsburgh Sleep Dairy (PghSD) will be used to assess sleep perceived quality. The PghSD is an instrument with separate components to be completed at bedtime and wake time. The following parameters are registered or assessed:
  Bedtime, wake time, sleep latency, wake after sleep onset, total sleep time, mode of awakening and ratings of sleep quality, mood, and alertness on wakening, as well as daytime information on naps, exercise, meals and caffeine, tobacco and medications use.
Change in psychological state: mental health | At baseline and until week 12
  General Health Questionnaire-28 (GHQ-28) will be used to assess psychological well-being and capture distress
  GHQ-28 gives an overall total score and 4 scores for 4 subscales:
  Somatic symptoms, Anxiety/insomnia, Social dysfunction, Severe depression. Higher scores indicate higher levels of distress
Measurement of changes in subjective sleep quality | At baseline and until week 12
  Changes in subjective sleep quality will be measured using the Karolinska sleepiness scale (KSS) two times per day (bed time) every week.

SECONDARY OUTCOMES:
Change in vertebral bone marrow fat fraction. | At baseline and until year 1
  This will be performed by using MR scanning sequences that specifically measure water and fat signals then calculate the respective content.
Changes in myokinins. | At baseline and until week 12
  Mass spectrometry will be performed on proteins obtained from muscle biopsies, microdialysis and serum. The generated peptides will be analysed using high resolution mass shot-gun mass spectrometry.
Changes in brain structure | At baseline and until week 12
  Both structural and functional brain changes associated with head-down bedrest will be examined by 3 Tesla MRI. Imaging sequence parameters will be selected to maximize sensitivity to effects of interest.
Change in pulse wave velocity in carotid and femoral arteries | At baseline and until year 1
  Change in pulse wave velocity in carotid and femoral arteries will be assessed by non-invasive ultrasound measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Billette de Villemeur, Principal Investigator — MEDES - Institut de Médecine et Physiologie Spatiale
Locations (1):
- MEDES-Institut de Médecine et Physiologie Spatiale, Toulouse, France, France